CLINICAL TRIAL: NCT05713357
Title: Repeated Endocardial Mapping for Efficacy Assessment After Catheter Ablation for Ischemic Ventricular Tachycardia
Acronym: REMAP-VT
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matevz Jan, Electrophysiology Specialist, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: VT remap
Record Dates: First submitted 2023-01-15; First posted 2023-02-06 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Cardiomyopathy; Ventricular Tachycardia
Keywords: Catheter Ablation; Repeated Mapping
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation — Endocardial catheter ablation

SUMMARY:
Patients with ischemic ventricular tachycardia (VT) are frequently treated with radiofrequency catheter ablation. The efficacy of catheter ablation is limited for various reasons; one of those being incomplete myocardial and inhomogenous scar tissue damage due to suboptimal ablation lesions.

The aim of our study is to reassess initially ablated endocardial areas in a repeated mapping procedure. Initial lesion parameters will be studied in areas with conduction recovery at repeated mapping procedure. Also, VT inducibility will be correlated to the extent and characteristics of areas with recovered conduction.

DETAILED DESCRIPTION:
Patients with ischemic ventricular tachycardia and implanted defibrillatior (ICD) will be sent to catheter ablation according to current guidelines (ESC and/or HRS). At the initial procedure the scar will be mapped with an ablation catheter and a high density catheter and all abnormal endocardial electrical potentials will be marked on a three-dimensional electro-anatomical (3DEAM) map; late potentials, local abnormal ventricular activity and decrement evoked electrical potentials. Afterwards, programed ventricular stimulation will be performed with an intent to induce sustained ventricular tachycardia. Imaging derived three-dimensional reconstructions of the ischemic scar will be used according to the operator's discretion.

All regions with abnormal endocardial electrical potentials will be ablated with an irrigated, contact force enabled catheter with a power setting of 30-50W. The aim during each energy delivery will be near-field electrical signal dissapearance or absence of myocardial capture at high energy local electrical stimulation. All ablated regions will be re-mapped during the same procedure with a high density mapping catheter. Additional ablation will be performed until all near-field electrical signals are be abolished.

The endpoint of each procedure will be absence of near-field electrical signals in the ablated areas and noninducibility of sustained ventricular tachycardia at the repeated programed ventricular stimulation.

After 1-3 months all patients will have a re-mapping procedure with a high density catheter. Programmed ventricular stimulation will be performed. If any sustained ventricular tachycardia will be induced or if any residual abnormal endocardial electrical potentials will be found in previously ablated regions, additional ablations will be performed with identical ablation settings and endpoints as in the initial procedure.

All areas previously ablated and with recovered electrical conduction will be identified, marked on the 3DEAM map and used for analysis with inclusion of ablation parameters and findings at the initial procedure and (non)inducibility of the sustained ventricular tachycardia at the repeat procedure.

Patients will be followed-up ICD interrogation at scheduled ambulatory visits or reports from emergency or other department using recorded electrocardiograms (ECG).

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease,
* sustained ventricular tachycardia,
* implanted (or scheduled for implantation) cardiac electrical device with ability to record and store intracardiac electrograms

Exclusion Criteria:

* nonischemic cardiomyopathy,
* need for epicardial access to the substrate for treatment of ventricular tachycardia,
* any severe acute organ damage beyond cardiomyopathy that could potentialy omit remapping procedure after 3 months,
* any terminal disease with expected survival of less than one year

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic cardiomyopathy with a clear indication to undergo catheter ablation for treatment of sustained ventricular tachycardia according to recognized and current guidelines (ESC and/or HRS).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Absence of electrical activity in previously ablated areas | 3 months
  Absent electrical activity in segments of the left ventricle ablated at initial procedure - assessed according to 17 segment model of the left ventricle, using three-dimensional electro-anatomic mapping system and high-density mapping tools.
  Absence of electrical activity in previously ablated segments will be regarded as a positive outcome.
  Presence of electrical activity will be regarded as recurrence of conduction and considered a negative outcome and a measure of procedural failure.
Inducibility of ventricular tachycardia at repeat procedure | 3 months
  Inability to induce ventricular tachycardia with programed stimulation at repeat procedure will be considered a positive outcome. Inducibility of ventricular tachycardia will be considered a negative outcome and a measure of procedural failure.

SECONDARY OUTCOMES:
Recurrence of ventricular tachycardia | 1 year
  Recurrence of ventricular tachycardia detected with an implanted electrical device (ICD, CRT-D of ILR) during the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Matevž Jan, MD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; ESC Scientific Document Group. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J. 2015 Nov 1;36(41):2793-2867. doi: 10.1093/eurheartj/ehv316. Epub 2015 Aug 29. No abstract available. PMID 26320108
- [Background] Aktas MK, Younis A, Zareba W, Kutyifa V, Klein H, Daubert JP, Estes M, McNitt S, Polonsky B, Goldenberg I. Survival After Implantable Cardioverter-Defibrillator Shocks. J Am Coll Cardiol. 2021 May 25;77(20):2453-2462. doi: 10.1016/j.jacc.2021.03.329. PMID 34016257
- [Background] Pedersen CT, Kay GN, Kalman J, Borggrefe M, Della-Bella P, Dickfeld T, Dorian P, Huikuri H, Kim YH, Knight B, Marchlinski F, Ross D, Sacher F, Sapp J, Shivkumar K, Soejima K, Tada H, Alexander ME, Triedman JK, Yamada T, Kirchhof P, Lip GY, Kuck KH, Mont L, Haines D, Indik J, Dimarco J, Exner D, Iesaka Y, Savelieva I; EP-Europace,UK. EHRA/HRS/APHRS expert consensus on ventricular arrhythmias. Heart Rhythm. 2014 Oct;11(10):e166-96. doi: 10.1016/j.hrthm.2014.07.024. Epub 2014 Aug 30. No abstract available. PMID 25179489
- [Background] Fernandez-Armenta J, Soto-Iglesias D, Silva E, Penela D, Jauregui B, Linhart M, Bisbal F, Acosta J, Fernandez M, Borras R, Villuendas R, Cano L, Guasch E, Mont L, Berruezo A. Safety and Outcomes of Ventricular Tachycardia Substrate Ablation During Sinus Rhythm: A Prospective Multicenter Registry. JACC Clin Electrophysiol. 2020 Oct 26;6(11):1435-1448. doi: 10.1016/j.jacep.2020.07.028. PMID 33121673
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Result] Oloriz T, Baratto F, Trevisi N, Barbaro M, Bisceglia C, D'Angelo G, Yamase M, Paglino G, Radinovic A, Della Bella P. Defining the Outcome of Ventricular Tachycardia Ablation: Timing and Value of Programmed Ventricular Stimulation. Circ Arrhythm Electrophysiol. 2018 Mar;11(3):e005602. doi: 10.1161/CIRCEP.117.005602. PMID 29545359